CLINICAL TRIAL: NCT00822861
Title: A Single Center, Open Label, Stepwise, Dose Profiling Study to Evaluate the Efficacy and Safety of Four Dose Regimens of Inhaled TPI ASM8 in Patients With Allergic Asthma
Brief Title: Efficacy and Safety of Four Escalating Dose Regimens of TPI ASM8 in Patients With Allergic Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Syntara (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPI ASM8-206
Record Dates: First submitted 2009-01-13; First posted 2009-01-15 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — TPI ASM8

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dose level No.1 (Experimental): TPI ASM8 1 mg BID
  Interventions: Drug: TPI ASM8
- Dose level No.2 (Experimental): TPI ASM8 2 mg BID
  Interventions: Drug: TPI ASM8
- Dose level No.3 (Experimental): TPI ASM8 4mg BID
  Interventions: Drug: TPI ASM8
- Dose level No.4 (Experimental): TPI ASM8 8 mg Die
  Interventions: Drug: TPI ASM8

INTERVENTIONS:
Drug: TPI ASM8 — 4 mg/mL, 1 mg BID for 4 days
  Other Names: ASM8
  Arms: Dose level No.1
Drug: TPI ASM8 — 4 mg/mL, 2 mg BID for 4 days
  Other Names: ASM8
  Arms: Dose level No.2
Drug: TPI ASM8 — 4 mg/mL, 4 mg BID for 4 days
  Other Names: ASM8
  Arms: Dose level No.3
Drug: TPI ASM8 — 4 mg/mL, 8 mg OD for 4 days
  Other Names: ASM8
  Arms: Dose level No.4

SUMMARY:
During this proposed clinical trial, the investigators intend to evaluate the pharmacodynamic anti-inflammatory properties and safety of TPI ASM8, by investigating the effect on sputum eosinophils and the airway responses during an allergen challenge at different dose levels.

DETAILED DESCRIPTION:
The early and late asthmatic response were both significantly attenuated by the highest dose of ASM8. The methacholine challenge and other parameters (ECP, mRNA knockdown on CCR3 and B-Chain of IL-3-Il-5 and GMCSF were attenuated by ASM8.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 to 65 years of age
* Generally good health; steroid naïve (or who have not taken inhaled/oral corticosteroid within last month) mild to moderate, stable, allergic asthma as defined by ATS criteria
* History of episodic wheeze and shortness of breath
* Forced expiratory volume in one second (FEV1) at baseline ≥ 70% of the predicted value
* Able to comprehend and follow all required study procedures; willing and able to sign an informed consent form.

Exclusion Criteria:

* Significant acute or chronic medical or psychiatric illness
* Known coagulopathy, worsening of asthma or respiratory infection in the preceding 6 weeks
* Use of inhaled or oral corticosteroids within the last 30 days, or need for antihistamines within 72 hours of each allergen or methacholine challenge, immunosuppressives, nonsteroidal anti-inflammatory drugs, or anticoagulants (intermittent doses of short-acting β2-agonist are allowed).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-04; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Sputum eosinophils (%) on Day 4 versus Screening for each dose level. | 7 and 24 hrs post-allergen challenge

SECONDARY OUTCOMES:
Safety and tolerability. | Throughout the study
Plasma and sputum pharmacokinetic profile at the two highest dose levels. | Dose level 3 and 4

CONTACTS AND LOCATIONS:
Overall Officials: Rene Pageau, B.Pharm M.Sc, Study Director — Topigen Pharmaceuticals Inc.
Locations (1):
- McMaster University, Hamilton, Ontario, Canada